CLINICAL TRIAL: NCT06266013
Title: Influence of an Inspiratory Muscle Fatigue Protocol on Older Adults on Respiratory Muscle Strength, Muscle Oxygen Saturation, and Functional Capacity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sierra Varona SL (Other)
Collaborators: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 009
Record Dates: First submitted 2024-01-24; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: the outcome assessor will not know in which group is each participant, and the investigator will receive the data without knowing which data is from which group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group (Experimental): The EG (experimental group) will perform the diaphragmatic fatigue protocol using a specific inspiratory endurance test, in which volunteers, one-on-one, and in a single session, will breathe against submaximal inspiratory loads equivalent to 60% of their MIP (Maximum Inspiratory Pressure) through a threshold valve device. The participants will follow a free pattern of breathing until they are unable to establish flow during at least 3 maximum inspiratory efforts.
  Interventions: Other: inspiratory muscle training
- control group (No Intervention): they will not receive any intervention. Just sit and wait the same amount of time that the intervention and the activation group needs to finish their protocol (around 10 minutes)
- activation group (Active Comparator): The activation group will perform the protocol of 2 sets of 30 repetitions at 15% of their MIP, one-on-one, and in a single session, breathing against submaximal inspiratory loads using a threshold valve device. The participants will follow a free pattern of breathing until complete the protocol.
  Interventions: Other: inspiratory muscle training

INTERVENTIONS:
Other: inspiratory muscle training — The subjects will perform deep inspirations against a threshold device with varying resistances to observe the effect on the diaphragm and the musculature of the lower limbs.
  Other Names: inspiratory muscle fatigue
  Arms: activation group; intervention group

SUMMARY:
Respiratory muscle training represents an effective method increasingly utilized in both sports and healthcare domains, employing various devices, among which threshold devices are prominent. The aim of this study is to determine the relationship between diaphragmatic fatigue and muscular strength in upper and lower limbs, in both healthy and pathological subjects, as well as the association between such fatigue and other variables, including maximal inspiratory pressure, functionality and muscle tissue oxygen levels.

According to our hypothesis, the execution of a protocol inducing diaphragmatic fatigue in older adults could influence muscular strength, cardiorespiratory function, exercise capacity, and muscle tissue oxygenation.

In this study, subjects will be divided into three groups: the experimental group , the activation group and the control group.

Measurements of variables, such as maximal inspiratory pressure, peripheral muscle tissue oxygen levels, diaphragmatic strength (ultrasound image) and functional capacity, will be conducted.

DETAILED DESCRIPTION:
this is a randomized control trial. The experimental group (EG) will perform the diaphragmatic fatigue protocol using a specific inspiratory endurance test, in which volunteers, one-on-one, and in a single session, will breathe against submaximal inspiratory loads equivalent to 60% of their Maximum Inspiratory Pressure (MIP) through a threshold valve device. The participants will follow a free pattern of breathing until they are unable to establish flow during at least 3 maximum inspiratory efforts.

The activation group (AG) will perform the protocol of 2 sets of 30 repetitions at 15% of their MIP, one-on-one, and in a single session, using a threshold valve device.

The control group will do a seat and wait.

The interventions will be supervised by a physiotherapist. The primary outcomes will be

* Muscle oxygen saturation (SmO2) will be assessed using a near infrared spectroscopy device, immediately before intervention and immediately after intervention
* Functional mobility will be assessed using the Timed Up and Go Test (TUG) immediately before intervention and immediately after intervention
* Respiratory muscle strength will be assessed using a respiratory pressure meter or manometer designed, and with ultrasound image measuring the cross sectional area of the diaphragm at 8-9th rib level and speed of contraction with a deep and fast inspiratory manoeuver. This will be done immediately before intervention and immediately after intervention
* Functional capacity will be assessed using the Five sit to Stand Test (5STS) Immediately before intervention and immediately after intervention.

ELIGIBILITY:
Inclusion Criteria:

* • Being over 60 years old.

  * Physical independence in terms of gait and transfers

Exclusion Criteria:

* Having any pathology that prevents the performance of physical activity.

  * Subjects with impaired cognitive abilities.
  * Subjects with tympanic perforation or middle-inner ear pathology.
  * Subjects with pulmonary hypertension, decompensated heart or respiratory failure.
  * Subjects who have undergone lower limb surgery within the past 12 months.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-02-14 (Estimated); Primary Completion 2024-02-19 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Muscle oxygen saturation (SmO2) | Pre intervention and post intervention
  is a physiological assessment that measures the saturation level of oxygen in muscles during exercise. it utilizes near-infrared spectroscopy (NIRS) technology, often in the form of a device that includes sensors placed on the skin above the target muscles. During the exercise, the NIRS device continuously measures the levels of oxygenated and deoxygenated hemoglobin in the muscles. The measures will be expressed in %.
Functional mobility | Pre intervention and post intervention
  It will be assessed using the Timed Up and Go Test (TUG). The Time Up and Go (TUG) test is a widely used clinical assessment to evaluate mobility, functional mobility, and fall risk in individuals, particularly the elderly:
  Procedure:
  The individual starts by sitting in a standard armchair or chair with a backrest.
  Upon the command "Go," the person stands up from the chair. The individual walks a distance of 3 meters (about 10 feet) as quickly and safely as possible.
  Once they reach a marker or a designated spot, they turn around. The person walks back to the chair and sits down.
  The measures will be expressed in seconds.
Respiratory muscle strength | Pre intervention and post intervention
  It will be assessed using a MicroRPM® (MicroMedical, UK).The MicroRPM® is likely a respiratory pressure meter or manometer designed for measuring respiratory muscle strength. It typically includes a mouthpiece connected to a pressure sensor, and the device measures the force or pressure generated during respiratory maneuvers.
  Procedure:
  Preparation: The individual undergoing the test will be instructed on the procedure. They may sit or stand comfortably during the assessment.
  Mouthpiece Placement: The individual will be asked to place the mouthpiece securely in their mouth, ensuring a tight seal to prevent air leakage.
  Respiratory Maneuvers:
  Maximum Inspiratory Pressure (MIP): The person will be instructed to take a maximal deep breath in, and then exhale to residual volume. After that, they will be asked to inhale forcefully against the resistance provided by the MicroRPM®. This measures the strength of the inspiratory muscles.
  The measures will be expressed in cmH2O.
Diaphragmatic thickness and thickening fraction | Pre intervention and post intervention
  Diaphragmatic thickness and thickening fraction The linear array probe with a frequency of 3.0-10 megahertz (MHz) is placed perpendicularly to chest wall close to the mid-axillary line which is between the 8th and 10th intercostal space. The thickness of diaphragm is measured at the end of expiration and maximum inspiration for three times and the average values were recorded.
  The measures will be expressed in centimeters.
Functional capacity | Pre intervention and post intervention
  It will be assessed using the Five sit to Stand Test (5STS). It is a functional capacity assessment that measures an individual's ability to transition from a seated to a standing position.he individual starts in a seated position on a chair with a standardized height (typically armless and around knee height).
  The feet are flat on the floor, shoulder-width apart.On the command to start, the person stands up from the chair completely and then returns to the seated position. This process is repeated four more times, making a total of five sit-to-stand transitions.
  The measures will be expressed in seconds.
Diaphragm movement curve | Pre intervention and post intervention
  The convex array probe with a frequency of 1.5-4.6 MHz is placed below the midclavicular line of the right costal margin in longitudinal scanning plane. The liver was used as an inspection window, and the probe was pointed toward the cephalic side. The ultrasound bundle is perpendicular to the posterior third of the right diaphragm. M-mode ultrasound is used to record the diaphragmatic movement curve during quiet breathing (QB) and deep breathing (DB).
  The measures will be expressed in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: arturo ladriñan, Principal Investigator — Universidad Europea de Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ladrinan-Maestro A, Sanchez-Infante J, Martin-Vera D, Sanchez-Sierra A. Influence of an inspiratory muscle fatigue protocol on older adults on respiratory muscle strength, muscle oxygen saturation, and functional capacity: a randomized controlled trial. BMC Geriatr. 2024 Dec 19;24(1):1015. doi: 10.1186/s12877-024-05610-0. PMID 39702081